CLINICAL TRIAL: NCT02387541
Title: Effects of Total Knee Replacement on Early Postoperative Cognitive Function in Elderly Patients
Acronym: POCD
Status: Completed | Type: Observational
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NZ10145
Record Dates: First submitted 2015-03-06; First posted 2015-03-13 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2015-03

CONDITIONS: Perioperative Complications
Keywords: Postoperative cognitive dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To investigate the effects of total knee replacement is harmful to Postoperative cognitive dysfunction

DETAILED DESCRIPTION:
Postoperative cognitive dysfunction (POCD) is reported to occur after major surgery in elderly patients. They may especially experience problems in the weeks and months after surgery. Recent studies vary greatly in methods of evaluation and diagnosis of POCD, and the pathogenic mechanisms are still unclear. The investigators evaluated a large uniform cohort of elderly patients in a standardized approach after total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥65 years;
* ASA I or Ⅱ;
* total knee replacement

Exclusion Criteria:

* Mini Mental State Examination [MMSE] score too low.
* Parkinson or other neurological disease causing functional impairment.
* Patients with a history of alcohol abuse (≥35 U per week) or daily use of anxiolytics were also excluded, as well as those with severe hearing or visual impairment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: We included 96 ASA I or Ⅱ patients aged ≥65 years performed total knee replacement under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Effects of operation on early postoperative cognitive function in elderly patients | up to 7days postoperatively

SECONDARY OUTCOMES:
Postoperative cognitive dysfunction (POCD) was defined by Mini-Mental State Examination (MMSE) score | up to 7days postoperatively

OTHER OUTCOMES:
serum concentration of inflammatory cytokine | The blood samples were reserved before anesthesia induction and 24h after surgery
  The blood samples were reserved before anesthesia induction and 24h after surgery for detecting the concentrations of IL-1, IL-6, and IL-10 by enzyme-linked immunosorbent assay (ELISA).